CLINICAL TRIAL: NCT02418962
Title: Phase 1, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Safety and Immunogenicity of Direct Venous Inoculation of a Radiation-attenuated Plasmodium Falciparum Sporozoite Vaccine (PfSPZ Vaccine) in Equatoguinean Adults
Brief Title: Safety and Immunogenicity of Direct Venous Inoculation of a Radiation-attenuated PfSPZ Vaccine in Equatoguinean Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Government of Equatorial Guinea (Other Government); Hospital Universitario La Paz (Other); Marathon Oil Corporation (Industry); Noble Oil Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EGSPZV1
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: PfSPZ Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (pilot group) (Experimental): Group 1 will be comprised of 3 volunteers who will be vaccinated first before the rest for demonstration of safety. The safety volunteers will receive 2 escalating doses of PfSPZ vaccine at a two week interval, 1.35x10^5 and 2.7x10^5 PfSPZ.
  Interventions: Biological: PfSPZ Vaccine
- Group 2 (Experimental): The second group of 14 - 20 volunteers will receive three vaccinations of 2.7x10^5 PfSPZ Vaccine that will be given at 0, 8 and 16 weeks
  Interventions: Biological: PfSPZ Vaccine
- Group 3 (Placebo Comparator): The third group of 7 - 10 volunteers will act as control group for group 2 and will receive three injections of normal saline at 0, 8 and 16 weeks respectively.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, metabolically active, non-replicating (live, radiation attenuated) cryopreserved Plasmodium falciparum sporozoites vaccine
  Arms: Group 1 (pilot group); Group 2
Other: Normal Saline — 0.9% Sodium chloride solution for injection
  Arms: Group 3

SUMMARY:
This is a single center, randomized, placebo-controlled, double-blind trial to assess the safety and immunogenicity of PfSPZ Vaccine administered by direct venous inoculation (DVI).

The study to be conducted in Baney District, Bioko Island, Equatorial Guinea (EG), will be to establish whether three doses of the higher regimen - three doses of 2.7x10^5 PfSPZ of the PfSPZ Vaccine administered at 8 week intervals - is as well-tolerated and efficacious in malaria exposed African adults as the five dose regimens. Specifically, the trial will address the following objectives: is the three dose regimen:

1. Safe and well tolerated in Equatoguinean (EG) adults.
2. As immunogenic in EG adults as is the five-dose regimen of 1.35x10^5 PfSPZ in Tanzanian and U.S. adults or as three-, four- and five-dose regimens of 2.7x10^5 PfSPZ being tested in Tanzanian, Malian and U.S. adults.

In addition, as an exploratory objective, the volunteers in the EG trial will be followed longitudinally to measure the incidence of malaria during the initial six months following immunization, providing a preliminary assessment of efficacy.

DETAILED DESCRIPTION:
This is a single center, Phase 1, randomized, double-blind, placebo-controlled trial. Thirty-three healthy male volunteers, aged 18 to 35 years will be recruited into three groups. The first group will be comprised of 3 volunteers who will be vaccinated first before the rest for demonstration of safety. The safety volunteers will receive 2 escalating doses of PfSPZ vaccine at a two week interval, 1.35x10^5 and 2.7x10^5 PfSPZ. The second group of 14 - 20 volunteers will receive three vaccinations of 2.7x10^5 PfSPZ that will be given at 0, 8 and 16 weeks (in the Tanzania trial, volunteers will receive a five dose regimen at 0, 4, 8, 12 and 18 weeks). The third group of 7 - 10 volunteers will act as control group for group 2 and will receive three injections of normal saline at 0, 8 and 16 weeks respectively.

Volunteers in groups 2 and 3 will only be injected when the Safety Monitoring Committee (SMC) provides clearance based on the results from the sentinel 3 volunteers (group 1). For groups 2 and 3, five volunteers will be vaccinated with the first dose before the remaining volunteers are vaccinated on a subsequent day.

The control volunteers will help better assess the occurrence of adverse events compared to background disease patterns that occur in this tropical area. The decision to dose escalate in group 1 and to immunize a larger number of volunteers in group 2 in Bioko will be made with full knowledge of all safety data generated in other ongoing trials where the PfSPZ Vaccine is being tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy literate male aged between 18 - 35 years
* Good health status based on history and clinical examination.
* Long term (at least two year) or permanent residence in the city of Baney or community of Rebola, Bioko Island, Equatorial Guinea
* Free from malaria parasitaemia by blood smear at screening
* Not suffering from any chronic illness including HIV/AIDS.
* Able and willing to come for complete one year follow up.
* Answered correctly 10 out 10 questions demonstrating their understanding of study and study procedures.
* Written informed consent.
* Volunteer agrees to inform study doctor and agrees to release medical information concerning contra-indications for participation in the study.
* Living with a third party who will contact the study team, if there is any alteration of consciousness during the first six months of the study.
* Willingness to be attended by a study clinician and take all necessary medications prescribed during study period.
* Availability through mobile phone 24 hours during the whole study period.
* Agreement not to participate in another study during the study period.
* Agreement not to donate blood during the study period.
* Willingness to attend all study visits.
* Willingness to undergo HIV, hepatitis B and hepatitis C tests.

Exclusion Criteria:

* Plans to travel outside the Bioko, Equatorial Guinea in first nine months of the study.
* Previous receipt of an investigational malaria vaccine or participation in a malaria drug study.
* History of arrhythmias or prolonged QT-interval or other cardiac disease.
* History of drug or alcohol abuse interfering with normal social function.
* A history of psychiatric disease.
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period.
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, blood, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers.
* History of diabetes mellitus or cancer.
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.
* Clinically significant abnormalities in electrocardiogram (ECG) at screening.
* Body Mass Index (BMI) below 18 or above 30 kg/m2.
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis or electrolytes.
* Positive HIV, hepatitis B virus or hepatitis C virus tests.
* Participation in any other clinical study within 30 days prior to the onset of the study or during the study period.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Study team employees and their immediate family relatives.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia.
* Risk factor for clinically active tuberculosis + positive tuberculin skin test (TST)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | Until 28 days after each vaccination
  Occurrence of solicited adverse events during a 7-day surveillance period after vaccination (day of vaccination and study days 1, 2, 3, 4, 5 and 6). Occurrence of unsolicited adverse events during a 28-day surveillance period after each vaccination.
Number of serious adverse events | From first vaccination upto 50 weeks
  Occurrence of serious adverse events during the study period.
Number of Pf infections | From first vaccination upto 50 weeks
  Occurrence of Pf infection of vaccine type detected at any point after the first vaccination (retrospectively determined).

SECONDARY OUTCOMES:
Antibody titers to PfCSP, PfLSA-1, PfEXP-1 and PfMSP-5 by ELISA | Before each vaccination, at 2 and 4 weeks after 1st and 2nd vaccinations (groups 2 and 3) and at 2, 4, 8, and 24 weeks after the last vaccination.
  Antibody titers to PfCSP, PfLSA-1, PfEXP-1 and PfMSP-5 by ELISA, and their functional activity to block invasion of hepatocytes at screening, before each vaccination, at 2 and 4 weeks after the first and second vaccinations (groups 2 and 3) and at 2, 4, 8, and 24 weeks after the last vaccination.
Antibody titers to whole Pf sporozoite by Immunofluorescence (IFA) | Before each vaccination, 2 and 4 weeks after each vaccination, and at 8, and 24 weeks after the last vaccination.
  Antibody titers to whole Pf sporozoite by Immunofluorescence (IFA) and their functional activity to block invasion of hepatocytes at screening, before each vaccination, 2 and 4 weeks after each vaccination, and at 8, and 24 weeks after the last vaccination.
Cellular immune responses | Screening and at 2 and 24 weeks after the last vaccination
  Cellular immune responses to the whole PfSPZ and synthetic peptides from selected Pf pre-erythrocytic antigens by ELISPOT and Intracellular Cytokine Staining (ICS) at screening and at 2 and 24 weeks after the last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdulla, MD, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- La Paz Medical Center, Malabo, Equatorial Guinea

REFERENCES:
- [Derived] Olotu A, Urbano V, Hamad A, Eka M, Chemba M, Nyakarungu E, Raso J, Eburi E, Mandumbi DO, Hergott D, Maas CD, Ayekaba MO, Milang DN, Rivas MR, Schindler T, Embon OM, Ruben AJ, Saverino E, Abebe Y, Kc N, James ER, Murshedkar T, Manoj A, Chakravarty S, Li M, Adams M, Schwabe C, Segura JL, Daubenberger C, Tanner M, Richie TL, Billingsley PF, Lee Sim BK, Abdulla S, Hoffman SL. Advancing Global Health through Development and Clinical Trials Partnerships: A Randomized, Placebo-Controlled, Double-Blind Assessment of Safety, Tolerability, and Immunogenicity of PfSPZ Vaccine for Malaria in Healthy Equatoguinean Men. Am J Trop Med Hyg. 2018 Jan;98(1):308-318. doi: 10.4269/ajtmh.17-0449. Epub 2018 Jan 1. PMID 29141739